CLINICAL TRIAL: NCT06270316
Title: A Phase 1/2, Single Dose, Dose Ranging Study of Intravenous AAV5-GLA (AMT-191) in Adult Males With Classic Fabry Disease
Brief Title: Safety, PK/PD, and Exploratory Efficacy Study of AMT-191 in Classic Fabry Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UniQure Biopharma B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-AMT-191-01
Record Dates: First submitted 2023-12-19; First posted 2024-02-21 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Fabry Disease
Keywords: GLA; gene therapy; ERT; FD
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Ranging Cohort 1 (Experimental)
  Interventions: Drug: AMT-191
- Dose Ranging Cohort 2 (Experimental)
  Interventions: Drug: AMT-191
- Dose Ranging Cohort 3 (Experimental)
  Interventions: Drug: AMT-191

INTERVENTIONS:
Drug: AMT-191 — A recombinant serotype 5 based adeno-associated viral vector (AMT-191) for one-time intravenous (IV) administration will be investigated in this study. This recombinant AAV5-based vector contains a coding deoxyribonucleic acid (DNA) sequence for human α-galactosidase A.
  Delivery of AMT-191 to the systemic circulation is expected to result in a therapeutic effect by promoting the liver expression of the lysosomal enzyme GLA in plasma levels in patients with Fabry disease.

SUMMARY:
The main goals of this clinical study are to characterize safety and PK/PD of AMT-191 i.e. if drug doses used in the study are safe and tolerable and to understand how it acts in the body of people with Fabry disease.

DETAILED DESCRIPTION:
In Fabry disease, the enzyme α-galactosidase A is deficient. AMT-191 is an investigational gene therapy that encodes a recombinant serotype 5 based adeno-associated viral vector (rAAV5). AMT-191 is designed to target the liver for production of the enzyme α-galactosidase A (αGAL). AMT-191 is delivered via a single (one-time) intravenous (IV) infusion.

In this first-in-human study of AMT-191, two or more dose levels will be tested.

All eligible participants will receive AMT-191 at one of the dose levels; there is no placebo in this study. The starting dose level is decided based on accepted rules for dose translation from preclinical (animal) studies to humans. Subsequent dose cohort levels are decided based on the review of safety, tolerability, and PK/PD results by an Independent Data Monitoring Committee and in agreement with the Sponsor.

Participants will be monitored through study site visits, blood tests, imaging questionnaires, and other assessments as per the study protocols.

ELIGIBILITY:
Key Inclusion Criteria:

* Male of age ≥ 18 years and ≤50 years
* Confirmed clinical diagnosis of classic Fabry disease (FD) defined as:

  1. Absent or minimal αGAL A enzyme activity < 1% of mean normal measured in plasma regardless of variant status; OR
  2. α-galactosidase A (GLA) pathogenic or likely pathogenic variant associated with classic FD phenotype identified on molecular genetic testing with plasma αGLA A enzyme activity below lower bound of the reference range (as measured at trough enzyme replacement therapy [ERT] levels).
* eGFR ≥ 40 mL/min/1.73 m2
* Suboptimal response after at least 12 months of enzyme replacement therapy (ERT) treatment. Suboptimal response is defined as plasma lyso-Gb3 ≥ 2.3 nanograms per milliliter (ng/mL) at Screening and one or both of the following:
* Persistent moderate or severe neuropathic pain (intermittent or continuous) over a period of at least 3 months prior to consent
* Presence of gastrointestinal symptoms (abdominal cramping, constipation, or diarrhea), reported by the Participant as moderate or severe and that are either persistent or occurring two or more times over the 12 weeks prior to consent
* Weight ≤ 120 kilograms (kg)

Key Exclusion Criteria:

* Any allergic hypersensitivity reaction to ERT or infusion reaction in the 12 months prior to consent that was of severity grade 3 or above based on Common Terminology Criteria for Adverse Events (CTCAE v5.0) and required emergency intervention for hypertension/hypotension to stabilize blood pressure or hypoxia OR any other life-threatening complication.
* Proteinuria, with random urine protein/creatinine ratio (rUPCR) ≥1 mg/mg at Screening
* Current use of chaperone therapy such as migalastat (Galafold®)
* Malignancy within 5 years of Screening, except for basal or squamous cell carcinoma of the skin
* Presence of chronic, active, or latent infection with hepatitis B or C, human immunodeficiency virus (HIV), or tuberculosis (TB) as assessed at the screening visit
* Active or ongoing infection or any other significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, cardiovascular, hematological, GI, endocrine (such as diabetes mellitus with poor glycemic control), pulmonary, neurological, cerebral, or psychiatric disease, alcoholism, drug dependency, or any other psychological disorder that could, in the opinion of the Investigator, risk the safety of the Participant, or interfere with adherence to the protocol procedures or interpretation of results
* Evidence of any liver disease, including hepatitis, fibrosis, cirrhosis of the liver, neoplastic lesion, or any known medical condition that could impact the intended transduction of the vector and/or expression and activity of the protein
* History of kidney transplantation or currently on hemodialysis or peritoneal dialysis
* Uncontrolled hypertension, defined as systolic blood pressure >140 millimeters of mercury (mmHg) (inclusive) and/or diastolic blood pressure outside the range of 60 to 85 mmHg (inclusive) at Screening, confirmed on at least 2 repeated measurements
* Patients taking blood pressure medication to control blood pressure or proteinuria (eg, angiotensin-converting enzyme [ACE] inhibitors and angiotensin II receptor blockers [ARBs]) and have been titrated to a stable dose for at least 3 months prior to Screening are allowed in the study.
* Glycated hemoglobin (HbA1c) at Screening ≥7%
* Contraindication to systemic corticosteroid therapy or immunosuppressive therapy
* Chronic steroid use, defined as ≥ 3 months of oral corticosteroid use within the 12 months prior to Screening
* Screening laboratory values for renal and liver function that meet or exceed any of the following:

  1. Alanine transaminase (ALT) > 2 x upper limit of normal for the testing laboratory (ULN)
  2. Aspartate aminotransferase (AST) > 2 x ULN
  3. Total Bilirubin > 2 x ULN (except if this is caused by Gilbert disease)
  4. Alkaline phosphatase (ALP) > 2 x ULN
  5. Creatinine > 2 x ULN
* Screening laboratory values for hematologic and coagulation function that meet any of the following:

  1. Hemoglobin < lower limit of normal (LLN) (as per reference laboratory ranges)
  2. Platelet count < 150 x1000/μl
  3. International normalized ratio (INR) >1.1
  4. Soluble terminal complement complex (sC5b-9)>ULN
* Significant anatomical abnormalities on renal ultrasound such as the presence of only 1 kidney, significant differences in kidney sizes between the right and left kidneys >1.5 centimeters (about 0.59 inch), or presence of kidney cysts

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male of age ≥ 18 years and ≤ 50 years
Enrollment: 12 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of different dose levels of intravenously-administered AMT-191 in Participants with FD | 60 Months
Incidence of Treatment-Emergent Adverse Events (TEAE) | 60 Months

SECONDARY OUTCOMES:
Characterize the vector shedding of intravenously-administered AMT-191 | 60 Months
  Duration of vector deoxyribonucleic acid (DNA) shedding present in blood, saliva, feces, semen, and urine.

CONTACTS AND LOCATIONS:
Overall Officials: Arian Pano, MD, MPH, Study Director — Clinical Development and Progam Lead, uniQure Biopharma, B.V.
Locations (8):
- United States (8):
  - The Kirklin Clinic Of university of Alabama Birmingham Hospital, Birmingham, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - MHealth Fairview University of Minnesota Medical Center East Bank, Minneapolis, Minnesota
  - NYC Health + Hospitals/Metropolitan, New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Clinical and Translational Sciences Institute, Salt Lake City, Utah
  - Lysosomal & Rare Disorders Research and Treatment Center, Inc, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No